CLINICAL TRIAL: NCT03159351
Title: Repetitive Transcranial Magnetic Stimulation for Depression After Basal Ganglia Ischemic Stroke: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Antidepressant Effects of rTMS After Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-SJNK-005
Record Dates: First submitted 2017-05-01; First posted 2017-05-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active rTMS treatment (Experimental): received active rTMS treatment 20 times for 20 days
  Interventions: Device: active rTMS treatment
- sham rTMS treatment (Sham Comparator): received sham rTMS treatment 20 times for 20 days
  Interventions: Device: sham rTMS treatment

INTERVENTIONS:
Device: active rTMS treatment — active rTMS treatment protocol parameters: localization of left DLPFC: frequency=10 Hz, intensity=110% motor threshold(MT), times per train=200 seconds, trains=10, duration= 40 seconds, total times=20;localization of right DLPFC: frequency=1 Hz, intensity=100%MT, times per train=30 seconds, trains=10, duration= 10 seconds, total times=20.
  Arms: active rTMS treatment
Device: sham rTMS treatment — sham rTMS treatment protocol parameters: sham rTMS treatment in the localization of left DLPFC and right DLPFC for 30 minutes,total times=20.
  Arms: sham rTMS treatment

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled trial aims to assess the effectiveness of repetitive transcranial magnetic stimulation(rTMS) in treating depression after basal ganglia ischemic stroke and to examine whether such effects are related to restoration of white matter integrity.Sixty-six participants will be recruited from three centers and randomized with a 1:1 ratio to receive active rTMS treatment or sham rTMS treatment in addition to routine supportive treatments.The data of neuropsychological tests and MRI will be collected at 0, 2 and 4 weeks after the commencement of the treatment.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial aims to assess the effectiveness of rTMS in treating depression after basal ganglia ischemic stroke and to examine whether such effects are related to restoration of white matter integrity.Sixty-six participants will be recruited from three centers and randomized with a 1:1 ratio to receive active rTMS treatment or sham rTMS treatment in addition to routine supportive treatments.The data of neuropsychological tests and MRI will be collected at 0, 2 and 4 weeks after the commencement of the treatment.The primary outcome is the measurement of 24-item Hamilton Depression Rating Scale (HAMD-24) scores, and the secondary outcomes include diffusion tensor imaging (DTI) results and the results of neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA),Clinical Global Impressions scales(CGI), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire (MCMQ).

ELIGIBILITY:
Inclusion Criteria:

1. First-time ischemic stroke with clinical and MRI or CT findings of basal ganglia ischemic stroke and a diagnosis of depression due to stroke based on The Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) and The International Classification of Diseases-10 (ICD-10-CM code 293.83[F06.32]);
2. Aged 25-75 years with a recent (from 3 weeks to 3 months) ischemic stroke;
3. Clear signs of neurological deficits in the acute phase;
4. Clear consciousness;
5. Right-handedness.

Exclusion Criteria:

1. Aphasia or severe cognitive impairment, severe hearing impairment, or severe language comprehension deficits due to other causes;
2. Other cerebral diseases such as Parkinson's disease, encephalitis, dementia, multiple sclerosis, head injury, ect.;
3. Severe systemic disease or ongoing neoplasia;
4. Ongoing post-operative recovery;
5. Prior history of depressive disorders or major trauma within 1 year, severe depression or any other severe mental disorders;
6. Current or prior antidepressant use for any reason;
7. Addiction to drugs, alcohol or other substances;
8. Contraindications of MRI scan and rTMS treatment such as pacemaker implantation, a history of epilepsy, major head trauma, and seizures, ect;
9. Pregnant or breast-feeding women;
10. Participation in other clinical research projects;
11. Refusal to sign informed consent of this study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
response rate | baseline, 2nd and 4th week
  Compare the HAMD-24 scores from baseline to the end of the treatment.the response to treatment is defined as at least a 50% reduction of the HAMD-24 total score with a final HAMD-24 score below 9. The response rate is defined as the percentage of number of response.
remission rate | baseline, 2nd and 4th week
  Compare the HAMD-24 scores from baseline to the end of the treatment. The remission is defined as a reduction of the HAMD-24 total score by at least 50% from the baseline. The remission rate is defined as the percentage of number of remission.

SECONDARY OUTCOMES:
DTI results of FA | baseline and 4th week
  DTI parameters including the fractional anisotropy (FA), apparent diffusion coefficient (ADC), neural fiber number (NFN). Get the change of FA by Comparing the change of FA from baseline to the end of the treatment in each group.
DTI results of ADC | baseline and 4th week
  DTI parameters including the fractional anisotropy (FA), apparent diffusion coefficient (ADC), neural fiber number (NFN). Get the change of ADC by Comparing the change of ADC from baseline to the end of the treatment in each group.
DTI results of NFN | baseline and 4th week
  DTI parameters including the fractional anisotropy (FA), apparent diffusion coefficient (ADC), neural fiber number (NFN). Get the change of NFN by Comparing the change of NFN from baseline to the end of the treatment in each group.
Neuropsychological tests results of NIHSS | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of NIHSS by Comparing the change of NIHSS scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of ADLs | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of ADLs by Comparing the change of ADLs scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of MoCA | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of MoCA by Comparing the change of MoCA scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of ABC | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of ABC by Comparing the change of ABC scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of SSRS | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of SSRS by Comparing the change of SSRS scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of MCMQ | baseline and 4th week
  Neuropsychological tests including National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs), Montreal Cognitive Assessment (MoCA), Aphasia Battery in Chinese (ABC), Social Support Revalued Scale (SSRS) and Medical Coping Questionnaire score (MCMQ). Get the change of the result of MCMQ by Comparing the change of MCMQ scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of CGI | baseline and 4th week
  Neuropsychological tests including Clinical Global Impressions scales

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, Chen A, Zhu S, Yang L, Zhou J, Pan S, Shao M, Zhao L. Repetitive transcranial magnetic stimulation for depression after basal ganglia ischaemic stroke: protocol for a multicentre randomised double-blind placebo-controlled trial. BMJ Open. 2018 Feb 3;8(2):e018011. doi: 10.1136/bmjopen-2017-018011. PMID 29431126